CLINICAL TRIAL: NCT02477839
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Investigate the Efficacy and Safety of Lacosamide as Adjunctive Therapy in Subjects With Epilepsy >=1 Month to <4 Years of Age With Partial-Onset Seizures
Brief Title: Efficacy and Safety of Lacosamide as Adjunctive Therapy in Subjects ≥1 Month to <4 Years With Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP0967; 2013-000717-20 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2015-05-13; First posted 2015-06-23 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Epilepsy With Partial-onset Seizures
Keywords: Epilepsy; children; partial-onset seizures; lacosamide; LCM; pediatric
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lacosamide (Experimental): Lacosamide syrup 8 mg/kg/day to 12 mg/kg/day
  Interventions: Drug: Lacosamide
- Placebo (Placebo Comparator): Matching placebo syrup
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lacosamide — Active Substance: Lacosamide Pharmaceutical Form: Syrup Concentration: 10 mg/mL Route of Administration: oral
  Other Names: Vimpat; UCB Code: SPM 927; Abbreviated name: LCM
  Arms: Lacosamide
Other: Placebo — Active Substance: Placebo Pharmaceutical Form: Syrup Concentration: N/A Route of Administration: oral
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess the efficacy, safety and tolerability of lacosamide administered as add-on therapy with 1 to 3 anti-seizure medications. This trial is for children aged 1 month to less than 4 years with epilepsy who currently have uncontrolled partial-onset seizures.

DETAILED DESCRIPTION:
The trial consists of a 7-day Baseline Period, a 20-day Titration Period, a 7-day Maintenance Period, and a 12-day Transition Period for subjects who complete the study and choose to enter the extension study. Subjects who will not enter the extension study will continue after the Maintenance Period with a 16-day Taper Period followed by a 30-day Safety Follow-Up Period. The Taper Period and Safety Follow-Up are also applicable for subjects not eligible for continuation and therefore ending the study earlier.

If subjects meet the eligibility criteria, they will be randomized to receive either lacosamide 8 mg/kg/day to 12 mg/kg/day, or placebo during the Maintenance Phase. The dose of lacosamide will be titrated from 4 mg/kg/day at study start to maximum of 12 mg/kg/day at 4-day intervals of 1-2 mg/kg/day.

All subjects who complete the 20-day Titration Period will enter the 7-day Maintenance Period. No dose adjustment is allowed during the Maintenance Phase. The Treatment Phase is defined as the combined Titration and Maintenance Phases.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female from >=1 month (ie, 4 weeks after full term [37 weeks gestational age]) to <4 years of age
* Subject has a diagnosis of epilepsy with partial-onset seizures. The results of >=1 prior EEG and >=1 magnetic resonance imaging/computerized tomography scan should be consistent with this diagnosis
* Subject weighs >=4 kg to <30 kg at Visit 1
* Subject has experienced >=2 partial-onset seizures with or without secondary generalization during each consecutive 7-day period during the 2 weeks prior to Visit 1
* Subject has >=2 partial-onset seizures with or without secondary generalization during the End-of-Baseline video-EEG. Electrographic seizures are defined as recognizable ictal patterns on an EEG involving >=2 contiguous electrodes. The seizures are initiated as a unilateral or strongly asymmetric abnormal epileptiform discharge lasting a total of >10 seconds
* Subject is on a stable (concurrently or sequentially) dosage regimen of 1 to 3 AEDs. The dosage regimen of concomitant AED therapy must be kept constant for a period of >=2 weeks prior to Visit 1. A stable daily dosage regimen of a concomitant benzodiazepine (BZD) will be considered as a concomitant AED
* Vagus nerve stimulation (VNS) is allowed and will not be counted as a concomitant AED. The VNS device must have been implanted for >=6 months prior to Visit 1; device settings must be kept stable for >=2 weeks prior to Visit 1 and kept stable during the Baseline, Treatment, and Transition Periods. Use of the VNS device magnet is allowed
* Subject is an acceptable candidate for venipuncture

Exclusion Criteria:

* Subject has experienced febrile seizures exclusively. The occurrence of febrile seizures in addition to partial-onset seizures is not exclusionary
* Subject is on a ketogenic diet that has either changed within the 4 weeks prior to Visit 1 or is expected to change during the study
* Subject has creatinine clearance <30 mL/minute
* Subject has a clinically relevant ECG abnormality, in the opinion of the investigator (eg, second or third degree heart block at rest or a corrected QT interval [QTc] >=450 ms)
* Subject has a hemodynamically significant congenital heart disease
* Subject has an arrhythmic heart condition requiring medical therapy
* Subject has a known history of severe anaphylactic reaction secondary to medication intake or serious blood dyscrasias
* Subject has nonepileptic events that could be confused with seizures. Subjects may be included if epileptic events can be clearly distinguished and the frequency meets the study inclusion criteria
* Subject has a current diagnosis of Lennox-Gastaut syndrome, epilepsia partialis continua, primary generalized epilepsy, Dravet Syndrome, or seizures that are not of partial-onset origin
* Subject has a history of generalized convulsive status epilepticus <=2 months prior to Screening (Visit 1)
* Subject has been treated with felbamate and has experienced any serious toxicity issues (defined as liver failure, aplastic anemia) with this treatment. Subjects treated with felbamate for <12 months are excluded. Subjects treated with felbamate for >=12 months prior to Visit 1 and who have not experienced serious toxicity issues are eligible
* Subject has an acute or subacutely progressive central nervous system disease. Subject has epilepsy secondary to a progressing cerebral disease or any other progressively neurodegenerative disease (malignant brain tumor or Rasmussen Syndrome)
* Subject has a known cardiac sodium channelopathy, such as Brugada syndrome

Ages: 1 Month to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 255 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (88):
- United States (7):
  - Sp0967 638, Birmingham, Alabama
  - Sp0967 117, Tampa, Florida
  - Sp0967 115, Henderson, Nevada
  - Sp0967 120, Lebanon, New Hampshire
  - Sp0967 129, Dallas, Texas
  - Sp0967 630, San Antonio, Texas
  - Sp0967 643, San Antonio, Texas
- Sp0967 142, Córdoba, Argentina
- Brazil (4):
  - Sp0967 158, Passo Fundo
  - Sp0967 152, Porto Alegre
  - Sp0967 150, São Paulo
  - Sp0967 154, São Paulo
- Sp0967 310, Plovdiv, Bulgaria
- China (6):
  - Sp0967 530, Beijing
  - Sp0967 535, Changchun
  - Sp0967 532, Chongqing
  - Sp0967 536, Nanchang
  - Sp0967 531, Shanghai
  - Sp0967 537, Shenzhen
- Croatia (3):
  - Sp0967 613, Osijek
  - Sp0967 610, Rijeka
  - Sp0967 612, Zagreb
- Sp0967 320, Ostrava-Poruba, Czechia
- France (3):
  - Sp0967 349, Marseille
  - Sp0967 346, Rennes
  - Sp0967 344, Strasbourg
- Georgia (4):
  - Sp0967 620, Tbilisi
  - Sp0967 621, Tbilisi
  - Sp0967 622, Tbilisi
  - Sp0967 623, Tbilisi
- Sp0967 542, Athens, Greece
- Hungary (5):
  - Sp0967 361, Budapest
  - Sp0967 362, Budapest
  - Sp0967 363, Budapest
  - Sp0967 364, Budapest
  - Sp0967 368, Budapest
- Sp0967 374, Petah Tikva, Israel
- Italy (6):
  - Sp0967 397, Genova
  - Sp0967 398, Messina
  - Sp0967 381, Milan
  - Sp0967 700, Napoli
  - Sp0967 383, Roma
  - Sp0967 395, Roma
- Mexico (8):
  - Sp0967 694, Aguascalientes
  - Sp0967 561, Chihuahua City
  - Sp0967 569, Culiacán
  - Sp0967 693, Culiacán
  - Sp0967 563, Guadalajara
  - Sp0967 564, México
  - Sp0967 568, Monterrey
  - Sp0967 692, Monterrey
- Sp0967 650, Chisinau, Moldova
- Philippines (5):
  - Sp0967 720, Cebu
  - Sp0967 724, Cebu
  - Sp0967 721, Manila
  - Sp0967 723, Manila
  - Sp0967 727, Quezon City
- Sp0967 422, Krakow, Poland
- Sp0967 750, Lisbon, Portugal
- Romania (4):
  - Sp0967 581, Bucharest
  - Sp0967 582, Iași
  - Sp0967 573, Sibiu
  - Sp0967 577, Timișoara
- Russia (9):
  - Sp0967 454, Kemerovo
  - Sp0967 456, Nizhny Novgorod
  - Sp0967 452, Novosibirsk
  - Sp0967 453, Omsk
  - Sp0967 455, Perm
  - Sp0967 730, Smolensk
  - Sp0967 458, Tomsk
  - Sp0967 459, Ulyanovsk
  - Sp0967 450, Yekaterinburg
- Serbia (3):
  - Sp0967 461, Belgrade
  - Sp0967 464, Belgrade
  - Sp0967 463, Novi Sad
- Sp0967 474, Bratislava, Slovakia
- South Korea (2):
  - Sp0967 212, Seoul
  - Sp0967 215, Seoul
- Sp0967 224, Taipei, Taiwan
- Thailand (2):
  - Sp0967 237, Bangkok
  - Sp0967 235, Pathum Wan
- Ukraine (7):
  - Sp0967 602, Dnipro
  - Sp0967 609, Dnipro
  - Sp0967 681, Ivano-Frankivsk
  - Sp0967 600, Kiev
  - Sp0967 606, Kiev
  - Sp0967 682, Uzhhorod
  - Sp0967 603, Vinnytsia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in June 2015 and concluded in May 2020.
Pre-assignment Details: Completed study was defined as participants who had "Completed study participant" selected as status at termination. The total number of participants who completed the study comprises of those who completed the Transition Period and the ones that completed the Taper Period after completing the Maintenance Period.
  Participant Flow refers to the SS.
Groups:
- Placebo: Participants received matching placebo syrup.
- Lacosamide: Participants received lacosamide (LCM) syrup 8 mg/kg/day to 12 mg/kg/day.
Period: Overall Study
Arm/Group | Placebo | Lacosamide
Started | 127 | 128
Completed Transition Period | 124 | 117
Completed Taper After Maintenance | 0 | 1
Completed | 124 | 118
Not Completed | 3 | 10
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Participant had PGS during V6 | 0 | 1
Not completed — Parents decided to stop medication | 0 | 1
Not completed — Lack of tolerability | 0 | 1
Not completed — Exclusion criterion | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which consisted of all randomized study participants who took at least 1 dose of study medication.
Arm/Group | Placebo | Lacosamide | Total Title
Number analyzed (Participants) | 127 | 128 | 255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 127 | 128 | 255
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 26.1 (13.4) | 25.2 (13.6) | 25.6 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 57 | 109
  Male | 75 | 71 | 146
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 5 | 13 | 18
  Asian | 15 | 14 | 29
  Black | 0 | 2 | 2
  White | 101 | 94 | 195
  Other/Mixed | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Daily Frequency (ADF) of Electrographic Partial-onset Seizures From End-of-Baseline (EOB) Period Video-EEG to End-of-Maintenance (EOM) Period Video-EEG
Description: The change in ADF of electrographic partial-onset seizures as measured on the End-of-Maintenance Period video-electroencephalogram (EEG) compared to the End-of-Baseline Period video-EEG.
  Seizure frequency was analyzed using an analysis of covariance (ANCOVA) with terms for treatment, pooled randomized age stratum, pooled center, and Baseline seizure ADF. Seizure ADF was log transformed using the transformation of ln(X+1), where X is the seizure ADF. Baseline seizure ADF was log transformed.
  Least squares means were based on log-transformed data of the full ANCOVA model.
Time Frame: End-of-Baseline Period (Day -3 to Day 1) to End-of-Maintenance Period (Day 24 to Day 27)
Population: Full Analysis Set (FAS) included all study participants in the Safety Set (SS). The analysis consisted of all study participants in the FAS who had at least 48 hours of interpretable recordings during the EOB Period video-EEG and the EOM Period video-EEG.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Placebo (FAS): Participants received matching placebo syrup, forming the Full Analysis Set (FAS).
- Lacosamide (FAS): Participants received lacosamide (LCM) syrup 8 mg/kg/day to 12 mg/kg/day, forming the FAS.
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 120 | 116
percent change | 1.44 (0.06) | 1.40 (0.06)
Statistical Analysis 1: Comparison: Placebo (FAS) vs Lacosamide (FAS); Difference ratio in LS Mean was calculated as the exp [LSMLCM-LSMplacebo]; Test type: Other; ANCOVA; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [0.83 to 1.14]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Lacosamide (FAS); Percent reduction over placebo was estimated as 100 x (1-exp [LSMLCM-LSMPBO]); Test type: Other; p = 0.6895, ANCOVA; Percent reduction = 3.19, 95% CI 2-sided [-13.59 to 17.50]

2. Primary Outcome: Participant Withdrawals Due to Adverse Events (AEs) During the Study
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. An AE could, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study medication.
Time Frame: From the Baseline Period (Day -7) to the End of Study Visit (up to 93 days)
Population: The Safety Set (SS) included all randomized study participants who took at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (SS): Participants received matching placebo syrup, forming the Safety Set (SS).
- Lacosamide (SS): Participants received lacosamide (LCM) syrup 8 mg/kg/day to 12 mg/kg/day, forming the SS.
Arm/Group | Placebo (SS) | Lacosamide (SS)
Number analyzed (Participants) | 127 | 128
percentage of participants | 0 | 1.6

3. Primary Outcome: Percentage of Participants With Adverse Events Reported Spontaneously by the Participant's Parent(s) and/or Legal Representative(s)/Caregiver(s) (in Accordance With Local Regulation) or Observed by the Investigator
Description: as for outcome 2
Time Frame: From the Baseline Period (Day -7) to the End of Study Visit (up to 93 days)
Population: The Safety Set (SS) included all randomized study participants who took at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Lacosamide (SS)
Number analyzed (Participants) | 127 | 128
percentage of participants | 59.1 | 56.3

4. Secondary Outcome: Absolute Change in Average Daily Frequency (ADF) of Electrographic Partial-onset Seizures From End-of-Baseline (EOB) Period Video-EEG to End-of-Maintenance (EOM) Period Video-EEG
Description: The absolute change in ADF of electrographic partial-onset seizures as measured on the End-of-Maintenance Period video-EEG compared to the End-of-Baseline Period video-EEG.
Time Frame: End-of-Baseline Period (Day -3 to Day 1) to End-of-Maintenance Period (Day 24 to Day 27)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seizures per day
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 123 | 121
seizures per day | -4.7650 (18.0115) | -2.9427 (7.4938)

5. Secondary Outcome: Percent Change in Average Daily Frequency (ADF) of Electrographic Partial-onset Seizures From End-of-Baseline (EOB) Period Video-EEG to End-of-Maintenance (EOM) Period Video-EEG
Description: The percent change in ADF of electrographic partial-onset seizures as measured on the End-of-Maintenance Period video-EEG compared to the End-of-Baseline Period video-EEG.
Time Frame: End-of-Baseline Period (Day -3 to Day 1) to End-of-Maintenance Period (Day 24 to Day 27)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 122 | 121
percent change | -26.7927 (58.5564) | -32.3564 (65.0255)

6. Secondary Outcome: Percentage of Participants Who Achieved 'Seizure-free' Status From All Seizure Types During the End-of-Maintenance (EOM) Period Video-EEG
Description: A study participant was considered seizure-free from all seizures if the End-of-Maintenance (EOM) Period video-EEG had zero seizures reported from all seizure types (not just partial-onset seizures (POS)).
Time Frame: During the End-of-Maintenance Period (Day 24 to Day 27)
Population: Full Analysis Set (FAS) included all study participants in the Safety Set (SS). Percentages were based on the number of study participants in the FAS who completed at least 48 hours of interpretable video-EEG recordings during the EOM Period video-EEG.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 120 | 117
percentage of participants | 15.8 | 17.1

7. Secondary Outcome: Percentage of Participants Who Achieved 'Seizure-free' Status From Partial-onset Seizure Types Only During the End-of-Maintenance (EOM) Period Video-EEG
Description: A study participant was considered seizure free from partial-onset seizures (POS) if the End-of-Maintenance (EOM) Period video-EEG had zero POS reported.
Time Frame: During the End-of-Maintenance Period (Day 24 to Day 27)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 120 | 117
percentage of participants | 16.7 | 18.8

8. Secondary Outcome: Percentage of Participants Experiencing a >=25% to <50% Reduction in Average Daily Frequency (ADF) of Electrographic Partial-onset Seizures From End-of-Baseline (EOB) Period Video-EEG to End-of-Maintenance (EOM) Period Video-EEG
Description: A ≥25% to <50% response was defined as ≥25% to <50% reduction in ADF of electrographic partial-onset seizures (POS) from the End-of-Baseline (EOB) video-EEG to the End-of-Maintenance (EOM) video-EEG.
Time Frame: End-of-Baseline Period (Day -3 to Day 1) to End-of-Maintenance Period (Day 24 to Day 27)
Population: Full Analysis Set (FAS) included all study participants in the Safety Set (SS). Percentages were based on the number of study participants in the FAS who had at least 48 hours of interpretable recordings during the EOB Period video-EEG and the EOM Period video-EEG.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 120 | 116
percentage of participants | 18.3 | 18.1

9. Secondary Outcome: Percentage of Participants Experiencing a 50% to 75% Reduction in Average Daily Frequency (ADF) of Electrographic Partial-onset Seizures From End-of-Baseline (EOB) Period Video-EEG to End-of-Maintenance (EOM) Period Video-EEG
Description: A ≥50% to ≤75% response was defined as ≥50% to ≤75% reduction in ADF of electrographic partial-onset seizures (POS) from the End-of-Baseline (EOB) video-EEG to the End-of-Maintenance (EOM) video-EEG.
Time Frame: End-of-Baseline Period (Day -3 to Day 1) to End-of-Maintenance Period (Day 24 to Day 27)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 120 | 116
percentage of participants | 17.5 | 10.3

10. Secondary Outcome: Percentage of Participants Experiencing a >75% Reduction in Average Daily Frequency (ADF) of Electrographic Partial-onset Seizures From End-of-Baseline (EOB) Period Video-EEG to End-of-Maintenance (EOM) Period Video-EEG
Description: A >75% response was defined as >75% reduction in ADF of electrographic partial-onset seizures (POS) from the End-of-Baseline (EOB) video-EEG to the End-of-Maintenance (EOM) video-EEG.
Time Frame: End-of-Baseline Period (Day -3 to Day 1) to End-of-Maintenance Period (Day 24 to Day 27)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 120 | 116
percentage of participants | 20.0 | 31.0

11. Secondary Outcome: Percentage of Participants Experiencing no Change in Average Daily Frequency (ADF) of Electrographic Partial-onset Seizures (Between <25% Reduction and <25% Increase) From EOB Period Video-EEG to EOM Period Video-EEG
Description: No change was defined as between <25% reduction and <25% increase in ADF of electrographic partial-onset seizures (POS) from the End-of-Baseline (EOB) video-EEG to the End-of-Maintenance (EOM) video-EEG.
Time Frame: End-of-Baseline Period (Day -3 to Day 1) to End-of-Maintenance Period (Day 24 to Day 27)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 120 | 116
percentage of participants | 28.3 | 27.6

12. Secondary Outcome: Percentage of Participants Experiencing an Increase in Average Daily Frequency (ADF) of Electrographic Partial-onset Seizures of >=25% From End-of-Baseline (EOB) Period Video-EEG to End-of-Maintenance (EOM) Period Video-EEG
Description: An increase was defined as ≥25% increase in ADF of electrographic partial-onset seizures (POS) from the End-of-Baseline (EOB) video-EEG to the End-of-Maintenance (EOM) video-EEG.
Time Frame: End-of-Baseline Period (Day -3 to Day 1) to End-of-Maintenance Period (Day 24 to Day 27)
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 120 | 116
percentage of participants | 15.0 | 12.9

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the Titration Period (Day 1) to the End of Study Visit (up to 86 days)
Description: Treatment-emergent AEs (TEAEs) were defined as those events that start on or after the date of first study medication administration and within 30 days following the date of final study medication administration, or whose severity worsens within this time frame.
Arm/Group | Placebo (SS) | Lacosamide (SS)
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/128
Serious Adverse Events (participants affected / at risk) | 6/127 | 6/128
Other Adverse Events (participants affected / at risk) | 30/127 | 31/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=127) | Lacosamide (SS) (N=128)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 2 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=127) | Lacosamide (SS) (N=128)
Pyrexia (General disorders) | 15 (20) | 7 (9)
Irritability (General disorders) | 6 (6) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 13 (14) | 6 (6)
Somnolence (Nervous system disorders) | 5 (6) | 18 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT02477839/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT02477839/SAP_001.pdf